CLINICAL TRIAL: NCT05000411
Title: The Impact of Traditional Chinese Medicine, Compound Danshen Dropping Pills (CDDP) on the Post-myocardial Infarction Ventricular Remodeling: A Multicentre, Randomized, Double-blind, Placebo-controlled, Pilot Study
Brief Title: The Impact of Compound Danshen Dropping Pills (CDDP) on the Post-myocardial Infarction Ventricular Remodeling
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDDP
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Ventricular Remodeling; CDDP
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Compound Danshen Dropping Pills (CDDP)
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Compound Danshen Dropping Pills (CDDP) — The patients in this group are treated with 20 tablets of Compound Danshen Dropping Pills (CDDP) before primary Percutaneous Coronary Intervention (pPCI) and 10 tablets three times a day after pPCI.
  Arms: Experimental group
Drug: Placebo — The patients in this group take 20 tablets of placebo before primary Percutaneous Coronary Intervention (pPCI) and 10 tablets three times a day after pPCI .
  Arms: Control group

SUMMARY:
This study is designed to evaluate the efficacy and safety of compound Danshen dropping pills (CDDP) in improving ventricular remodeling and cardiac function after acute anterior wall ST-Elevation myocardial infarction(STEMI). 268 patients with acute anterior wall STEMI after primary Percutaneous Coronary Intervention (pPCI) are randomly assigned 1:1 to CDDP group(n=134) and control group(n=134) with follow-up of 24 weeks. Both groups are treated with standard therapy of STEMI, with the CDDP group administrating 20 tablets of CDDP before pPCI and 10 tablets three times a day after pPCI and the control group treated with placebo at the same time. The primary endpoint is 24-week echocardiographic including left ventricle ejection fraction (LVEF) , left ventricular end-diastolic volume index (LVEDVI) and left ventricular end-systolic volume index (LVESVI).The secondary endpoint is the change in N terminal pro-B-type natriuretic peptide（NT-proBNP ）level, arrhythmia and cardiovascular events (death, cardiac arrest or cardiopulmonary resuscitation, hospitalization due to heart failure or angina pectoris).

DETAILED DESCRIPTION:
Background: Progressive ventricular remodeling after acute anterior wall myocardial infarction（MI）is an important factor in the occurrence and death of heart failure. Angiotensin converting enzyme inhibitors and beta-blockers can ameliorate post-MI ventricular remodeling, but high-dose therapy can't be tolerable because of hemodynamic instability in the early stage of acute mycardial infarction（AMI）. It is known that traditional Chinese medicine, compound Danshen dropping pills (CDDP) exerts protective effect on microcirculatory disturbance caused by ischemia-reperfusion injury and improves energy metabolism after acute myocardial ischemia. Experimental studies have shown CDDP may attenuate ventricular remodeling after myocardial infarction.

Methods：This study is designed to evaluate the efficacy and safety of CDDP in improving ventricular remodeling and cardiac function after acute anterior wall ST-Elevation MI(STEMI). 268 patients with acute anterior wall STEMI after primary Percutaneous Coronary Intervention (pPCI) are randomly assigned 1:1 to CDDP group(n=134) and control group(n=134) with follow-up of 24 weeks. Both groups are treated with standard therapy of STEMI, with the CDDP group administrating 20 tablets of CDDP before pPCI and 10 tablets three times a day after pPCI and the control group treated with placebo at the same time. The primary endpoint is 24-week echocardiographic including left ventricle ejection fraction (LVEF) , left ventricular end-diastolic volume index (LVEDVI) and left ventricular end-systolic volume index (LVESVI).The secondary endpoint is the change in N terminal pro-B-type natriuretic peptide（NT-proBNP） level, arrhythmia and cardiovascular events (death, cardiac arrest or cardiopulmonary resuscitation, hospitalization due to heart failure or angina pectoris).

Discussion：This is the first prospective study that will demonstrate the impact of CDDP on ventricular remodeling and cardiac function in patients treated with pPCI for a first acute anterior wall STEMI .This study may provide novel insights of Traditional Chinese Medicine , CDDP to improve ventricular remodeling.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, gender unlimited;
2. According to the guidelines for diagnosis and treatment of acute ST segment elevation myocardial infarction (2019), patients with acute anterior ST segment elevation myocardial infarction were diagnosed;
3. Patients with primary acute myocardial infarction;
4. Patients who completed PCI reperfusion treatment within 12 hours after the onset of the disease;
5. Patients categorized as Classes I, II or III according to Killip classification on admission;
6. Subjects participated in the study voluntarily and signed informed consent.

Exclusion Criteria:

1. Patients with previous cardiac insufficiency caused by other diseases (valvular heart disease, congenital heart disease, pericardial disease, arrhythmia, other non cardiac causes);
2. The patients underwent coronary artery bypass graft（CABG） within 12 weeks;
3. Patients undergoing cardiac resynchronization;
4. Patients with left ventricular outflow tract obstruction;
5. Patients with myocarditis;
6. Patients with uncontrolled severe arrhythmia;
7. Patients with aortic aneurysm;
8. Patients with serious liver, kidney, blood system, mental disease or systemic disease;
9. Significant liver and kidney dysfunction (ALT > 2.0 times the upper limit of normal value; creatinine > 1.5 times the upper limit of normal value);
10. Patients with serum potassium > 5.5mmol/l;
11. Uncontrolled hypertension (higher than 180 / 110mmhg);
12. Pregnant or lactating women;
13. Patients allergic to compound Danshen Dropping Pills; 1
14. Patients participating in clinical studies of other drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-08-25 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
ultrasonic cardiogram：left ventricle ejection fraction (LVEF) | Week 24
  LVEF refers to the percentage of stroke output to left ventricular end-diastolic volume and it can be examined by ultrasonic cardiogram.
ultrasonic cardiogram：left ventricular end-diastolic volume index (LVEDVI) | Week 24
  LVEDVI（ml/m2）=left ventricular end-diastolic volume（ml）/body surface area（m2）. It can be examined by ultrasonic cardiogram.
ultrasonic cardiogram：left ventricular end-systolic volume index (LVESVI) | Week 24
  LVESVI（ml/m2）=left ventricular end-systolic volume（ml）/body surface area（m2）. It can be examined by ultrasonic cardiogram.

SECONDARY OUTCOMES:
N terminal pro-B-type natriuretic peptide（NT-proBNP ）decline level | Day 0/ Day 3/ Day 7/ Week 4/ Week 24/ Week 48
  N terminal pro-B-type natriuretic peptide（NT-proBNP ）is obtained by blood test.
Adverse cardiovascular events | Day 0 to Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wu YJ, Deng B, Wang SB, Qiao R, Zhang XW, Lu Y, Wang L, Gu SZ, Zhang YQ, Li KQ, Yu ZL, Wu LX, Zhao SB, Zhou SL, Yang Y, Wang LS. Effects of Compound Danshen Dripping Pills on Ventricular Remodeling and Cardiac Function after Acute Anterior Wall ST-Segment Elevation Myocardial Infarction (CODE-AAMI): Protocol for a Randomized Placebo-Controlled Trial. Chin J Integr Med. 2023 Dec;29(12):1059-1065. doi: 10.1007/s11655-023-3648-6. Epub 2023 Sep 1. PMID 37656413